CLINICAL TRIAL: NCT04339348
Title: Comparative Safety and Efficacy of Vaginal Misoprostol Versus Lidocaine-prilocaine Cream in Reducing Pain During Levonorgestrel IUD Insertion in Women Delivered Only by Cesarean Deliveries
Brief Title: Comparative Safety and Efficacy of Vaginal Misoprostol Versus Lidocaine-prilocaine Cream in Levonorgestrel IUD Insertion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: misoprostol vs LP cream
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vaginal misoprostol (Experimental): vaginal misoprostol 200 mcg will be given 3 hours before LNG-IUD insertion plus vaginal inert placebo cream at the time of IUD insertion
  Interventions: Drug: vaginal misoprostol
- lidocaine prilocaine cream (Active Comparator): Lidocaine-prilocaine anesthetic cream will be placed on the cervix at the time of IUD insertion plus vaginal placebo will be given 3 hours before LNG-IUD insertion
  Interventions: Drug: Lidocaine-Prilocaine Topical cream
- placebo (Placebo Comparator): inert vaginal placebo cream will be placed on the cervix at the time of IUD insertion plus vaginal placebo tablet will be given 3 hours before LNG-IUD insertion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vaginal misoprostol — vaginal misoprostol 200 mcg will be given 3 hours before LNG-IUD insertion plus inert placebo cream vaginally at the time of LNG-IUD insertion
  Arms: vaginal misoprostol
Drug: Lidocaine-Prilocaine Topical cream — Lidocaine-Prilocaine cream will be applied on the cervix at the time of LNG-IUD insertion plus vaginal placebo tablet 3 hours before LNG-IUD insertion
  Arms: lidocaine prilocaine cream
Drug: placebo — inert placebo cream will be applied on the cervix at the time of LNG-IUD insertion plus vaginal placebo tablet 3 hours before LNG-IUD insertion
  Arms: placebo

SUMMARY:
the aim of the present study is to compare the safety and Efficacy of vaginal misoprostol versus Lidocaine-prilocaine cream in reducing pain during levonorgestrel IUD Insertion in women delivered only by cesarean deliveries

ELIGIBILITY:
Inclusion Criteria:

* women who delivered only by previous cesarean delivery and requesting LNG-IUD insertion

Exclusion Criteria:

* women who delivered vaginally, active vaginal or cervical infections and contraindications to IUD insertion or study drugs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
pain during LNG-IUD insertion | 5 minutes
  pain during LNG-IUD insertion evaluated by 10 cm visual analog scale where 0 denotes no pain and 10 denotes the worst imaginable pain

SECONDARY OUTCOMES:
duration of insertion | 5 minutes
  duration of LNG-IUD insertion from speculum in to speculum out

CONTACTS AND LOCATIONS:
Overall Officials: ahmed taher, MD, Study Director — Cairo University; sherif dahab, MD, Principal Investigator — Cairo University; tarek el husseiny, Principal Investigator — Cairo University
Locations (1):
- Ahmedsamy, Giza, Egypt